CLINICAL TRIAL: NCT01236339
Title: The GORE® VIATORR® TIPS Endoprosthesis Versus Large-Volume Paracentesis for the Treatment of Ascites in Patients With Portal Hypertension
Brief Title: Early TIPS for Ascites Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTR 10-03
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Ascites
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIPS (Experimental): TIPS with GORE® VIATORR® TIPS Endoprosthesis
  Interventions: Device: TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis
- LVP (Active Comparator): Large Volume Paracentesis
  *A subject may be crossed-over from large volume paracentesis to TIPS with GORE® VIATORR® TIPS Endoprosthesis if the subject has completed their six month study visit and has met the criteria for cross-over (LVP failure).
  Interventions: Procedure: LVP; Device: TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis for subjects who failed LVP and crossed over to TIPS per protocol

INTERVENTIONS:
Device: TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis — TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis
  Arms: TIPS
Procedure: LVP — Large Volume Paracentesis
  Arms: LVP
Device: TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis for subjects who failed LVP and crossed over to TIPS per protocol
  Arms: LVP

SUMMARY:
The purpose of this study is to demonstrate that TIPS with the GORE® VIATORR® TIPS Endoprosthesis improves transplant-free survival compared to LVP alone in patients who have cirrhosis of the liver with portal hypertension and difficult to treat ascites.

ELIGIBILITY:
Inclusion Criteria:

> Patient has cirrhosis of the liver with portal hypertension

> Patient has difficult to treat ascites

> Patient is 18 years or older and <70 years old at randomization

> Patient is willing and able to comply with all study protocol requirements, including specified follow-up and testing.

> Patient, or legal authorized representative, is willing to provide written informed consent prior to enrollment in the study.

Exclusion Criteria:

> Patient has more than 6 large volume paracenteses within 90 days prior to randomization

> Patient is contraindicated for TIPS placement

> Patient has had previous TIPS placement

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Boyer, MD, Principal Investigator — University of Arizona College of Medicine; Ziv Haskal, MD, Principal Investigator — University of Maryland
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Maryland-Baltimore, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- LVP (Large Volume Paracentesis): Large Volume Paracentesis
  *A subject may be crossed-over from large volume paracentesis to TIPS with GORE® VIATORR® TIPS Endoprosthesis if the subject has completed their six month study visit and has met the criteria for cross-over (LVP failure)
Period: Overall Study
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Started | 13 | 13
LVP Crossover to TIPS | 0 | 4 (ONLY patients failing LVP and meeting crossover according to protocol definition)
Completed | 2 | 0
Not Completed | 11 | 13
Not completed — Termination of study by sponsor | 11 | 13

BASELINE CHARACTERISTICS:
Population: Patients who have cirrhosis of the liver with portal hypertension and difficult to treat ascites
Groups:
- TIPS: TIPS with GORE® VIATORR® TIPS Endoprosthesis >
  > TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis: TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis
- Total: Total of all reporting groups
Arm/Group | TIPS | LVP (Large Volume Paracentesis) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (6.6) | 57.5 (8.0) | 58.0 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20
  Canada | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Transplant-free Survival
Description: Time from randomization to death from any cause prior to transplant. Subjects who undergo liver transplant will be censored at the time of transplant. Subjects without an event will be censored at the date of last follow-up.
  * Note: The outcome entered below is the number of participants who were either alive or had a liver transplant at time of study termination.
Time Frame: Through 24 months
Measure: Number; unit: participants
Groups:
- LVP (Large Volume Paracentesis): LVP: Large Volume Paracentesis
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 13
participants | 11 | 13

2. Secondary Outcome: Overall Survival
Description: Time from randomization to death from any cause. Subjects without an event will be censored at the date of last follow-up. >
  *Note: Outcome measure entered below is number of subjects alive at time of study termination.
Time Frame: Through 24 months
Measure: Number; unit: participants
Groups:
- TIPS: TIPS with GORE® VIATORR® TIPS Endoprosthesis>
  > TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis: TIPS procedure with the GORE® VIATORR® TIPS Endoprosthesis
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 13
participants | 11 | 13

3. Secondary Outcome: Time to Transplant
Description: Time from randomization to transplant. Subjects without an event will be censored at the date of last follow-up or date of death without transplant.
  *Note: Outcome measure entered is number of subjects who received a liver transplant at time of study termination.
Time Frame: Through 24 months
Measure: Number; unit: participants
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 13
participants | 1 | 1

4. Secondary Outcome: Frequency of Paracentesis
Description: Number of paracentesis post randomization
Time Frame: Through 24 months
Measure: Number; unit: Number of episodes
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 13
Number of episodes | 25 | 93

5. Secondary Outcome: Frequency of Hepatic Encephalopathy
Description: Number of episodes of West Haven grade 2 or greater
Time Frame: Through 24 months
Measure: Number; unit: Number of episodes
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 13
Number of episodes | 4 | 2

6. Secondary Outcome: Procedural Success
Description: Successful creation of a VIATORR(R) device lined portosystemic shunt spanning a hepatic vein and intrahepatic branch of the portal vein
  *Note: Control (LVP) arm includes only subjects who crossed over to TIPS
Time Frame: Time of TIPS Procedure (within 2 weeks of enrollment for TIPS arm, at least 6 months after enrollment for Control arm crossover participants)
Measure: Number; unit: participants
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 4
participants | 12 | 4

7. Secondary Outcome: Liver Disease Complications (Adverse Events)
Description: Overall frequency and component frequencies. Complications will include hepatic encephalopathy, hepatic hydrothorax, hepatoma, hepatorenal syndrome (Type 1 or Type 2), hyponatremia (<130mEq / L), spontaneous bacterial peritonitis, and variceal bleeding.
Time Frame: Through 24 months
Measure: Number; unit: participants
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Number analyzed (Participants) | 13 | 13
participants
  Total Subjects with Liver Disease Complication | 5 | 4
  Subjects with Variceal Bleeding | 0 | 0
  Subjects with Hepatic Hydrothorax | 2 | 1
  Subjects with Hepatoma | 0 | 1
  Subjects with Hepatorenal Syndrome Type 1 | 0 | 0
  Subjects with Hepatorenal Syndrome Type II | 0 | 1
  Subjects with Hyponatremia | 1 | 1
  Subjects with Spontaneous Bacterial Peritonitis | 0 | 0
  Subjects with Hepatic Encephalopathy | 3 | 1

ADVERSE EVENTS:
Arm/Group | TIPS | LVP (Large Volume Paracentesis)
Serious Adverse Events (participants affected / at risk) | 6/13 | 2/13
Other Adverse Events (participants affected / at risk) | 3/13 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIPS (N=13) | LVP (Large Volume Paracentesis) (N=13)
Erosive esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Liver failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIPS (N=13) | LVP (Large Volume Paracentesis) (N=13)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)

LIMITATIONS AND CAVEATS:
Early termination due to very low enrollment.No subjects completed 24 month follow-up,sample size too small for adequate statistical analysis.Collected Adverse Events limited to hospitalizations and Liver Disease Complications as defined in protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites.